CLINICAL TRIAL: NCT01306019
Title: Lentiviral Gene Transfer for Treatment of Children Older Than 2 Years of Age With X-Linked Severe Combined Immunodeficiency
Brief Title: Lentiviral Gene Transfer for Treatment of Children Older Than Two Years of Age With X-Linked Severe Combined Immunodeficiency (XSCID)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110007; 11-I-0007
Record Dates: First submitted 2011-02-26; First posted 2011-03-01 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-06

CONDITIONS: X-linked Severe Combined Immunodeficiency (XSCID)
Keywords: T cell, B cell, NK cell; Gene Transfer; Peripheral Blood Stem Cells; Common Gamma Chain (gamma c); Immune Reconstitution
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases | interventions — Busulfan; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cohort a (Other): First 8 Patients Treated
  Interventions: Biological: Ex vivo culture and transduction of the patient's autologous CD34+ HSC with lentivirus vector VSV-G pseudotyped CL20- 4i-EF1alpha-hgammac-OPT vector; Drug: Busulfan; Drug: Palifermin
- cohort b (Other): Patients 9 and Beyond
  Interventions: Biological: Ex vivo culture and transduction of the patient's autologous CD34+ HSC with lentivirus vector VSV-G pseudotyped CL20- 4i-EF1alpha-hgammac-OPT vector; Drug: Busulfan; Drug: Palifermin

INTERVENTIONS:
Biological: Ex vivo culture and transduction of the patient's autologous CD34+ HSC with lentivirus vector VSV-G pseudotyped CL20- 4i-EF1alpha-hgammac-OPT vector — Transduced cell product administered intravenously over approximately 30 minutes by authorized licensed personnel consistent with NIH Clinical Center Department of Transfusion Medicine's standard operating procedures for cellular products.
Drug: Busulfan — 3mg/kg per day with drug levels obtained on Day -3. Busulfan dose on day -2 will be adjusted (if busulfan AUC result is available) to achieve targeted busulfan AUC 4500 min*umol/L/day. If the result is not available in time to adjust, then proceed to give the standard 3mg/kg on the second day
Drug: Palifermin — Mucositis prophylaxis commenced- Infusion of keratinocyte growth factor (palifermin) at 60 mcg/kg/day before (Days -6 to Day -4) administration of busulfan and (Days +1 to +3) post-busulfan administration

SUMMARY:
This is a Phase I/II non-randomized clinical trial of ex vivo hematopoietic stem cell (HSC) gene transfer treatment for X-linked severe combined immunodeficiency (XSCID, also known as SCID-X1) using a self-inactivating lentiviral vector incorporating additional features to improve safety and performance. The study will treat 35 patients with XSCID who are between 2 and 50 years of age and who have clinically significant impairment of immunity. Patients will receive a total busulfan dose of approximately 6 mg/kg/body weight (target busulfan Area Under Curve is 4500 min*micromol/L/day) delivered as 3mg/kg body weight on day 1 and dose adjusted on day 2 (if busulfan AUC result is available) to achieve the target dose, to condition their bone marrow, and this will be followed by a single infusion of autologous transduced CD34+HSC. Patients will then be followed to evaluate engraftment, expansion, and function of gene corrected lymphocytes that arise from the transplant; to evaluate improvement in laboratory measures of immune function; to evaluate any clinical benefit that accrues from the treatment; and to evaluate the safety of this treatment. The primary endpoint of the study with respect to these outcomes will be at 2 years, though data relevant to these measures will be collected at intervals throughout the study and during the longer follow-up period of at least 15 years recommended by the Food and Drug Administration (FDA) Guidance "Long Term Follow-Up After Administration of Human Gene Therapy Products" https://www.fda.gov/media/113768/download for patients

participating in gene transfer clinical trials.

XSCID results from defects in the IL2RGgene encoding the common gamma chain (yc) shared by receptors for Interleukin 2 (IL-2), IL-4, IL-7, IL-9, IL-15 and IL-21. At birth XSCID patients generally lack or have a severe deficiency of T-lymphocytes and NK cells, while their B- lymphocytes are normal in number but are severely deficient in function, failing to make essential antibodies. The severe deficiency form of XSCID is fatal in infancy without intervention to restore some level of immune function. The best current therapy is a T-lymphocyte-depleted bone marrow transplant from an HLA tissue typing matched sibling, and with this type of donor it is not required to administer chemotherapy or radiation conditioning of the patient's marrow to achieve excellent engraftment and immune correction of an XSCID patient. However, the great majority of patients with XSCID lack a matched sibling donor, and in these patients the standard of care is to perform a transplant of T- lymphocyte depleted bone marrow from a parent. This type of transplant is called haploidentical because in general a parent will be only half- matched by HLA tissue typing to the affected child. Whether or not any conditioning is used, haploidentical transplant for XSCID has a significantly poorer prognosis than a matched sibling donor transplant. Following haploidentical transplant, XSCID patients are observed to achieve a wide range of partial immune reconstitution and that reconstitution can wane over time in some patients. That subset of XSCID patients who either fail to engraft, fail to achieve adequate immune reconstitution, or lose immune function over time suffer from recurrent viral, bacterial and fungal infections, problems with allo- or autoimmunity, impaired pulmonary function and/or significant growth failure.

We propose to offer gene transfer treatment to XSCID patients^3 >= 2 years of age who have clinically significant defects of immunity despite prior haploidentical hematopoietic stem cell transplant, and who lack an HLA-matched sibling donor. Our current gene transfer treatment protocol can be regarded as a salvage/rescue protocol.

Prior successful retroviral gene transfer treatment instead of bone marrow transplant (BMT) in Paris and London for 20 infants with XSCID has provided proof of principle for efficacy. However, a major safety concern is the occurrence of 5 cases of leukemia at 3-5 years after treatment triggered in part by vector insertional mutagenesis activation of LMO2 and other DNA regulatory genes by the strong enhancer present in the long-terminal repeat (LTR) of the Moloney Leukemia Virus (MLV)- based vector.

Furthermore, previous studies of gene transfer treatment of older XSCID patients with MLV- based vectors demonstrated the additional problem of failure of adequate expansion of gene corrected T- lymphocytes to the very high levels seen in infants. To reduce or eliminate this leukemia risk, and possibly enhance performance sufficiently to achieve benefit in older XSCID patients, we have generated a lentivector with improved safety and performance features. We have generated a self-inactivating (SIN) lentiviral vector that is devoid of all viral transcription elements; that contains a short form of the human elongation factor 1a (EF1a) internal promoter to expres...

DETAILED DESCRIPTION:
This is a non-randomized clinical trial of gene transfer using a self-inactivating, insulated, lentiviral gene transfer vector to treat 35 patients with X-linked severe combined immunodeficiency (XSCID, also called SCID-X1) who are between 2 and 50 years of age; who do not have a tissue matched sibling who can donate bone marrow for a transplant; who may have failed to obtain sufficient benefit from a previous half-tissue matched bone marrow transplant; and who have clinically significant impairment of immunity. A patient s own precursor cells (also called blood stem cells) that give rise in the marrow to blood and immune cells will have been or will be collected from the patient s blood or bone marrow. A patient will not proceed to gene transfer treatment in this protocol until there are at least 3 million blood stem cells per kilogram body weight collected from the patient. At the NIH the patient blood stem cells will be cells collected previously under NIH protocol 94-1-0073 or collected on this protocol. In most cases the harvested blood stem cells are put into frozen storage before use in this protocol. When the patient enrolled in this protocol has the required number of blood stem cells harvested, then the patient s blood stem cells will be grown in tissue culture and exposed to the lentiviral gene transfer vector containing the corrective gene. These gene-corrected blood stem cells will be administered through the patient s vein. To increase engraftment of the corrected blood stem cells, patients will receive a chemotherapy drug called busulfan at a total dose of 6 mg/kilogram body weight (3 mg/kilogram body weight/daily) for two days before the gene transfer treatment. The busulfan dose to be used in this study is a little more than one-third the dose used in many standard bone marrow transplants. Patients will also be given another drug called palifermin that helps prevent the main side effect from the busulfan, which is a type of inflammation of the mouth, stomach and bowels called mucositis. After the gene transfer treatment, patients will be monitored to see if the treatment is safe and whether their immune system improves. Patients will be followed at frequent intervals for the first 2 years, and less frequently thereafter so that the effectiveness in restoration of immune function and the safety of the treatment can be evaluated.

XSCID is a genetic disease caused by defects in common gamma chain, a protein found at the surface of immune cells called lymphocytes and is necessary to their growth and function. XSCID patients cannot make T-lymphocytes necessary to fight infections, and their B-cells fail to make essential antibodies. Without normal T- and B-lymphocyte function patients develop fatal infections in infancy unless they receive a bone marrow transplant from a healthy donor. The best type of transplant is from a tissue matched healthy brother or sister, but most XSCID patients do not have a tissue-matched sibling and are treated with a transplant from a parent who is only half- matched by tissue typing. While a half-matched transplant from a parent can be lifesaving for an infant with XSCID, a subset of patients fails to achieve sufficient long lasting restoration of immunity to prevent infections and other chronic problems. Trials of gene transfer treatments using mouse retrovirus vectors for infants with XSCID have been performed and have demonstrated that this type of gene transfer can be an alternate approach for significantly restoring immunity to infants with XSCID. However, among the 18 infants with XSCID benefiting long-term from the gene transfer treatment, 5 developed Tlymphocyte leukemia and 1 died of this leukemia. Furthermore, when older children with XSCID were treated with gene transfer, the restoration of immunity was much less than seen in the infants. These observations of gene transfer treatments using mouse retrovirus vectors to treat infants and older patients with XSCID suggests that safer and more effective vectors were needed, and that there also may be a need to give chemotherapy or other method of conditioning to increase engraftment in the marrow of the gene corrected blood stem cells. Our data and other published studies suggest that lentivectors that are derived from the human immunodeficiency virus and have the properties of our highly modified vector called CL20-4i-EF1 - h >=c-OPT have a reduced interaction with nearby genes and therefore less of a tendency to activate genes that may lead to cancer formation. Also, this type of lentivector may work better at getting into blood stem cells.

The purpose of this study is to evaluate the safety and effectiveness of the lentiviral gene transfer treatment at restoring immune function to XSCID patients who are 2 to 50 years of age, and have significant impairment of immunity. Early evidence for effectiveness will be defined by appearance and expansion in the circulation of the patient s own gene corrected T-lymphocytes with a functional >=c gene and improved laboratory measures of immune function. The primary endpoint for efficacy will be at 2 years after treatment and will include these laboratory parameters plus evidence for clinical benefit. Evidence for safety will focus on the maintenance of a diversity of gene marked cells and no occurrence of abnormal patterns of production of blood cells or any leukemia or other cancer. The primary study endpoints for all laboratory and clinical measures of efficacy and safety will occur at 2 years after gene transfer treatment. However, data collection regarding efficacy will occur at frequent intervals during the 2 years leading up to the endpoint analysis, and long-term safety and efficacy evaluation will continue at intervals during the long-term follow-up period recommended by the United States FDA for patients participating in gene transfer treatment studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* A proven mutation in the common gamma chain gene as defined by direct sequencing of patient DNA
* No available HLA matched sibling donor as determined before enrollment. (HLA typing will be performed prior to enrollment)
* Must be between 2 and 50 years of age and weigh greater than or equal to 10 kg
* If previously transplanted, must be greater than or equal to 18 months post HSCT
* Expected survival of at least 120 days.
* Participants of reproductive potential must agree to consistently use highly effective contraception throughout study participation and for at least 2 years post-treatment. Acceptable forms of contraception are:

  --For males: Condoms or other contraception with partner.
* Documented to be negative for HIV infection by genome PCR
* The patient must be judged by the primary evaluating physician to have a suitable family and social situation consistent with ability to comply with protocol procedures and the long-term follow-up requirements.
* Medical lab data (historical) of severe B cell dysfunction (low or absent IgG levels, failed immune response to vaccines); OR demonstrated requirement for intravenous gamma globulin (IVIG) (significant drop over 3 to 6 weeks between peak and trough IgG levels).
* Must be willing to have blood and tissue samples stored IN ADDITION, patients must satisfy the following Laboratory Criteria AND Clinical Criteria

Laboratory Criteria: (greater than or equal to 1 must be present)

I. CD4+ lymphocytes: absolute number less than or equal to 50 percent of the lower limit of normal (LLN)

II. CD4+ CD45RA+ lymphocytes: absolute number less than or equal to 50 percent of the LLN OR T-cell receptor excision circles (TRECs) less than or equal to 5 percent of normal for age.

III. Memory B Cells: absolute number less than or equal to 50 percent of LLN

IV. Serum IgM<normal for age

V. NK cells: absolute number less than or equal to 50 percent of LLN

VI. Lymphocyte proliferative response to each of 2 mitogens, phytohemagglutinin (PHA) and concanavalin A (ConA), is <= 25 percent compared with a normal control.

VII. Molecular spectratype analysis- absent or very oligoclonal (1-3 dominant peaks) in greater than or equal to 6 of the 24 VBeta T-cell receptor families.

Clinical Criteria: (greater than or equal to 1 must be present):

I. Infections (not including molluscum, warts or mucocutaneous candidiasis; see vii and viii below):

Three significant new or chronic active infections during the 2 years preceding evaluation for enrollment, with each infection accounting for one criteria.

Infections are defined as an objective sign of infection (fever greater than 38.3 degrees C [101 degrees F] or neutrophilia or pain/redness/swelling or radiologic/ultrasound imaging evidence or typical lesion or histology or new severe diarrhea or cough with sputum production). In addition to one or more of these signs/symptoms of possible infection, there also must be at least 1 of the following criteria as evidence of the attending physician s intent to treat a significant infection (a. and b.) or objective evidence for a specific pathogen causing the infection (c.)

1. Treatment (not prophylaxis) with systemic antibacterial, antifungal or antiviral antibiotics greater than or equal to 14 days

   OR
2. Hospitalization of any duration for infection

   OR
3. Isolation of a bacteria, fungus, or virus from biopsy, skin lesion, blood, nasal washing, bronchoscopy, cerebrospinal fluid or stool likely to be an etiologic agent of infection

II. Chronic pulmonary disease as defined by:

1. Bronchiectasis by x-ray computerized tomography

   OR
2. Pulmonary function test (PFT) evidence for restrictive or obstructive disease that is 60 percent of Predicted for Age

   OR
3. Pulse oximetry 94 percent in room air (if patient is too young to comply with performance of PFTs).

III. Gastrointestinal enteropathy:

1. Diarrhea-watery stools greater than or equal to 3 times per day (of at least 3 months duration that is not a result of infection as defined in criterion above)

   OR
2. Endoscopic evidence (gross and histologic) for enteropathy (endoscopy will only be performed if medically indicated)

   OR
3. Other evidence of enteropathy or bacterial overgrowth syndrome: including malabsorption of fat-soluble vitamin(s), abnormal D-xylose absorption, abnormal hydrogen breath test, evidence of protein losing enteropathy (for example increasingly high or frequent dosing of intravenous gamma globulin supplement required to maintain blood IgG level).

IV. Poor nutrition: Requires G-tube or intravenous feeding supplement to maintain weight or nutrition.

V. Auto- or allo-immunity: Examples must include objective physical findings that include, but are not limited to any one of alopecia, severe rashes, uveitis, joint pain with redness or swelling or limitation of movement that is not a result of infection, lupus-like lesions, and granulomas (Does not include auto- or allo-immune enteropathy which is criterion iii). Where possible and appropriate, diagnosis will be supported by histopathology or other diagnostic modality.

VI. Failure to grow in height: less than or equal to 3rd percentile for age

VII. Skin molluscum contagiosum OR warts (this criterion is satisfied if molluscum consists of 10 lesions or there are two or more lesions at each of two or more widely separated anatomic sites; or there are 3 warts at different anatomic sites at the same time; or the patient has both molluscum and warts)

VIII. Mucocutaneous candidiasis (chronic oral thrush or candida esophagitis or candida intertriginous infection or candida nail infections; must be culture positive to satisfy this criterion)

IX. Hypogammaglobulinemia: requires regular IgG supplementation

EXCLUSION CRITERIA:

* Any current or pre-existing hematologic malignancy
* Documented HIV-1 infection
* Documented active Hepatitis B infection
* Childhood malignancy (occurring before 18 years of age) in the patient or a first degree relative, or previously diagnosed known genotype of the subject conferring a predisposition to cancer (no DNA or other testing for cancer predisposition genes will be performed as part of the screen for this protocol)

Ages: 2 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09-25 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Early evidence for efficacy will be defined by appearance and expansion in the circulation of autologous transduced T-lymphocytes with functional gmama-c and improved laboratory measures of immune function in the interim evaluation of these para... | 1 year
  successful, partial successful or failure

SECONDARY OUTCOMES:
evidence for efficacy at 2 years after treatment will include these same laboratory parameters measured at the 2 year time point plus evidence for clinical benefit | 2 years
  maintenance of polyclonality of vector marking, the lack of emergence of a dominant gene marked clone in any hematopoietic lineage, and no occurrence of either hematologic dysplasia or any leukemia or other cancer resulting from the gene transfer

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The PI has yet to determine how IPD will be shared.

REFERENCES:
- [Background] Howe SJ, Mansour MR, Schwarzwaelder K, Bartholomae C, Hubank M, Kempski H, Brugman MH, Pike-Overzet K, Chatters SJ, de Ridder D, Gilmour KC, Adams S, Thornhill SI, Parsley KL, Staal FJ, Gale RE, Linch DC, Bayford J, Brown L, Quaye M, Kinnon C, Ancliff P, Webb DK, Schmidt M, von Kalle C, Gaspar HB, Thrasher AJ. Insertional mutagenesis combined with acquired somatic mutations causes leukemogenesis following gene therapy of SCID-X1 patients. J Clin Invest. 2008 Sep;118(9):3143-50. doi: 10.1172/JCI35798. PMID 18688286
- [Background] Kang EM, Choi U, Theobald N, Linton G, Long Priel DA, Kuhns D, Malech HL. Retrovirus gene therapy for X-linked chronic granulomatous disease can achieve stable long-term correction of oxidase activity in peripheral blood neutrophils. Blood. 2010 Jan 28;115(4):783-91. doi: 10.1182/blood-2009-05-222760. Epub 2009 Dec 1. PMID 19965657
- [Background] Cartier N, Hacein-Bey-Abina S, Bartholomae CC, Veres G, Schmidt M, Kutschera I, Vidaud M, Abel U, Dal-Cortivo L, Caccavelli L, Mahlaoui N, Kiermer V, Mittelstaedt D, Bellesme C, Lahlou N, Lefrere F, Blanche S, Audit M, Payen E, Leboulch P, l'Homme B, Bougneres P, Von Kalle C, Fischer A, Cavazzana-Calvo M, Aubourg P. Hematopoietic stem cell gene therapy with a lentiviral vector in X-linked adrenoleukodystrophy. Science. 2009 Nov 6;326(5954):818-23. doi: 10.1126/science.1171242. PMID 19892975
- [Derived] De Ravin SS, Liu S, Sweeney CL, Brault J, Whiting-Theobald N, Ma M, Liu T, Choi U, Lee J, O'Brien SA, Quackenbush P, Estwick T, Karra A, Docking E, Kwatemaa N, Guo S, Su L, Sun Z, Zhou S, Puck J, Cowan MJ, Notarangelo LD, Kang E, Malech HL, Wu X. Lentivector cryptic splicing mediates increase in CD34+ clones expressing truncated HMGA2 in human X-linked severe combined immunodeficiency. Nat Commun. 2022 Jun 28;13(1):3710. doi: 10.1038/s41467-022-31344-x. PMID 35764638
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-I-0007.html